CLINICAL TRIAL: NCT03776773
Title: Impact of Pollution on Allergic Rhinitis and Sleep Quality: the POLLAR Study
Acronym: POLLAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 38RC18.264
Record Dates: First submitted 2018-12-13; First posted 2018-12-17 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Sleep Apnea; Allergic Rhinitis; Allergic Asthma; Pollution Exposure; Pollution Related Respiratory Disorder
MeSH Terms: conditions — Sleep Apnea Syndromes; Rhinitis, Allergic

STUDY DESIGN:
Intervention Model Description: Prospective, open study comparing sleep quality in 2 different groups: AR patients and patients without AR during the pollen season and outside the pollen season.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- patients AR (+) and sleep apnea (+) (Active Comparator): Patients with AR and obstructive sleep apnea (OSA) will have sleep and pollution exposure recordings
  Interventions: Other: Pollution exposure
- AR (-) and sleep apnea (+) (Active Comparator): Patients without allergic rhinitis (+ sleep apnea) will have sleep and pollution exposure recordings
  Interventions: Other: Pollution exposure
- AR (+) and sleep apnea (-) (Active Comparator): Patients with allergic rhinitis but no sleep apnea will have sleep and pollution exposure recordings
  Interventions: Other: Pollution exposure
- AR (-) and sleep apnea (-) (Sham Comparator): Volunteers without allergic rhinitis and no sleep apnea will have sleep and pollution exposure recordings
  Interventions: Other: Pollution exposure

INTERVENTIONS:
Other: Pollution exposure — Pollution exposure and sleep data will be recorded by pollution sensor and polysomnography respectively. In order to compare the variations according to the pollinisation season and the allergic rhinitis status of the patients.

SUMMARY:
It has been demonstrated that allergic rhinitis (AR) reduces sleep quality by some components such as nasal obstruction. Pollution and allergen exposure worsening AR, sleep quality is deteriorated.

Sleep is associated to physical and mental health, alterations in sleep could explain the link between AR and work productivity diminution, impairment in daily activities or emotional problems.

However, interactions between air pollution, sleep and allergic diseases are insufficiently understood.

The main objective of this study is to determine the impact of pollution and pollens on sleep parameters.

DETAILED DESCRIPTION:
Over 150 million people have allergic rhinitis (AR) in Europe and around 30% have uncontrolled AR during allergen exposure. It has been demonstrated that AR reduces sleep quality by some components such as nasal obstruction. Pollution and allergen exposure worsening AR, sleep quality is deteriorated.

Sleep is associated to physical and mental health, alterations in sleep could explain the link between AR and work productivity diminution, impairment in daily activities or emotional problems.

However, interactions between air pollution, sleep and allergic diseases are insufficiently understood.

Moreover, the prevalence of OSA in patients with AR is higher than in subjects without AR. Nasal obstruction could explain the increased risk of OSA.

This prospective, open study will compare sleep quality in 2 different groups: AR patients and patients without AR during the pollen season and outside the pollen season.The main objective is to determine the impact of pollution and pollens on sleep parameters for subjects with AR

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years
* Be able to use an application on a personal smartphone
* Patient non treated for OSA
* Be legally able to give consent
* Person affiliated to social security

Exclusion Criteria:

- Being unable to understand, follow objectives and methods due to cognition or language problems Subjects listed in articles L1121-5 à L1121-8: Pregnant women, feeding and parturient; subject under administrative or judicial control, persons who are protected under the act.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2020-01-25 (Actual); Study Completion 2020-01-25 (Actual)

PRIMARY OUTCOMES:
Impact of pollution on sleep | 6 days
  Change in AHI according to the level of pollution particle matters and volatile organic compounds (VOCs)

SECONDARY OUTCOMES:
The impact of pollution and pollens on sleep quality in patients with AR. | 6 days
  Change in Pittsburgh score according to the level of pollution particle matters and volatile organic compounds (VOCs)
The impact of pollution on life quality | 6 days
  Change in EQ-5D score according to the level of pollution particle matters and volatile organic compounds (VOCs)
To analyze variations in medications and impact on sleep during the pollen season and outside the pollen season. | 6 days
  Change in number of medications (antiallergics and hypnotics) according to the level of pollution particle matters and volatile organic compounds (VOCs)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis PEPIN, Principal Investigator — University Hospital, Grenoble
Locations (1):
- CHU Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided